CLINICAL TRIAL: NCT05314387
Title: A Multicentre, Prospective Clinical Study Analysing Outcomes of Shoulder Arthroplasty With SMR TT Hybrid Glenoid With or Without SMR Cementless Finned Short Stem
Brief Title: S-11 SMR TT Hybrid Glenoid and Cementless Finned Short Stem
Status: Not yet recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: S-11
Record Dates: First submitted 2022-03-18; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Shoulder Arthritis; Shoulder Osteoarthritis; Arthrosis; Osteoarthritis; Rheumatoid Arthritis; Arthroplasty; Avascular Necrosis; Humeral Fractures; Cuff Tear Arthropathy
Keywords: Shoulder Joint; Shoulder Replacement; Arthritis with rotator cuff tear; Post traumatic fracture sequele
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis; Humeral Fractures; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- SMR TT Hybrid Glenoid without Cementless Finned Short Stem: Patients implanted with SMR TT Hybrid Glenoid without Cementless Finned Short Stem
  Interventions: Device: SMR TT Hybrid Glenoid without Cementless Finned Short Stem
- SMR TT Hybrid Glenoid with Cementless Finned Short Stem: Patients implanted with SMR TT Hybrid Glenoid with Cementless Finned Short Stem
  Interventions: Device: SMR TT Hybrid Glenoid with Cementless Finned Short Stem

INTERVENTIONS:
Device: SMR TT Hybrid Glenoid without Cementless Finned Short Stem — The subject SMR Hybrid Glenoid System and SMR cementless finned short stem is intended for both primary or revision anatomic and reverse shoulder joint replacement. The glenoid components when used as part of an anatomic shoulder replacement are intended for cemented fixation.
  Groups: SMR TT Hybrid Glenoid without Cementless Finned Short Stem
Device: SMR TT Hybrid Glenoid with Cementless Finned Short Stem — The subject SMR Hybrid Glenoid System and SMR cementless finned short stem is intended for both primary or revision anatomic and reverse shoulder joint replacement. The glenoid components when used as part of an anatomic shoulder replacement are intended for cemented fixation.
  The fins are intended to enhance press-fit fixation. The same proximal morse taper is used for coupling to the same humeral bodies in the SMR Shoulder System. The SMR finned short stem is intended for cementless fixation.
  Groups: SMR TT Hybrid Glenoid with Cementless Finned Short Stem

SUMMARY:
Post-market, prospective, non randomized, open label, multicentre, clinical study analysing outcomes of shoulder arthroplasty with SMR TT Hybrid Glenoid with or without SMR Cementless Finned Short Stem

ELIGIBILITY:
Inclusion Criteria:(Key)

* Both genders;
* Age ≥ 18 years old;
* Full skeletal maturity;
* Life expectancy over 5 years;
* Patient is requiring primary unilateral arthroplasty based on physical examination and medical history;
* Good bone quality evaluated by the Investigator and the intraoperative evaluation;
* A diagnosis in the target shoulder of one or more of the S-11 SMR TT Hybrid Glenoid and Cementless Finned Short Stem Version Sep 2021 2.0 Confidential Page11 following:

  1. Primary osteoarthritis;
  2. Secondary osteoarthritis;
  3. Post-traumatic arthritis;
  4. Rheumatoid arthritis;
  5. Avascular necrosis
  6. acute fractures of the humeral head that cannot be treated with other fracture fixation methods;
  7. cuff tear arthropathy (only in combination with CTA Heads);
  8. Glenoid arthrosis without excessive glenoid bone loss: A1, A2 and B1 according to Walch classification.

Exclusion Criteria (Key):

* Patient requiring revision shoulder arthroplasty;
* Osteoporosis with a history of non-traumatic fractures;
* Steroid injections within the previous 3 months;
* Contralateral shoulder replacement within the previous 3 months;
* Significant proven or suspicious infection of the target shoulder or any serious infectious disease before the study according to the Investigator;
* Significant neurological or musculoskeletal disorders that may compromise functional recovery;
* Not recovered axillary nerve palsy;
* Non functioning deltoid muscle;
* Known or suspicious hypersensitivity to the metal or other components and materials of the implant;
* Participation in any experimental drug/device study within the 6 months prior to the preoperative visit;
* Women of childbearing potential who are pregnant, nursing, or planning to become pregnant.

These are key eligibility criteria, other eligibility criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopedic Clinics
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients reaching a clinical progression from baseline to 24-month follow-up | 24 Months
  The primary endpoint consists of the proportion of patients reaching a clinical progression from baseline to 24-month follow-up measured as:
  * Constant score improvement of greater than 10;
  * Adjusted Constant score greater than or equal to 54.

SECONDARY OUTCOMES:
Measure American Shoulder and Elbow Surgeons Shoulder Score (ASES) | Baseline to 24 and 60 Months
  The ASES questionnaire is composed of both a physician-rated component and a patient-reported component. The patient questions focus on joint pain, instability, and activities of daily living. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Measure Oxford shoulder score | Baseline to 24 and 60 Months
  Oxford Shoulder Score (OSS) is a 12-item patient-reported PRO specifically designed and developed for assessing outcomes of shoulder surgery.
Measure Constant Score | Baseline to 24 and 60 Months
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient. The higher the score, the higher the quality of the function.
Measure Simple Shoulder Test | Baseline to 24 and 60 Months
  Simple Shoulder Test (SST) is a series of 12 "yes" or "no" questions the patient answers about the function of the involved shoulder. The answers to these questions provides a standardized way of recording the function of a shoulder before and after treatment. The difference between the shoulder function before treatment and after the recovery period is the effectiveness of the treatment.
Measure Patient Satisfaction | Baseline to 24 and 60 Months
  The satisfaction of the patients with regard to the effectiveness of the prosthetic treatment is graded on a scale from 1 to 5
Stability of the SMR TT hybrid glenoid component with or without SMR cementless finned short stem | Immediately postoperative to 24 Months
  Rate of symptomatic radiolucent lines, loosening and subsidence ≥2 mm
System conversion rate, intended as a conversion within the SMR system from anatomic to reverse | 24 Months
  The SMR shoulder system is a modular system and in case of evolution of the pathology it may be easily converted from one configuration to another.
Failure rate, intended as removal of the SMR TT hybrid glenoid component | Immediately postoperative to 24 Months
  A removal of the glenoid component is intended as a revision and a failure of the implant.
Failure rate, intended as removal of the SMR cementless finned short stem | Immediately postoperative to 24 Months
  A removal of the stem component is intended as a revision and a failure of the implant.
Incidence of device-related AE/SAE (ADE/SADE) | Immediately postoperative to 24 and 60 Months
  Device Related Adverse Events/Serious Adverse Events, device deficiencies, malfunctions and use errors at all follow-up time points
Survival rate (Kaplan-Meier) | 60 Months

IPD SHARING:
Plan to Share IPD: No